CLINICAL TRIAL: NCT06666101
Title: Immunomodulatory Effects of Polyunsaturated ω-3 Fatty Acids in Old Patients With Polyvascular Disease: a Double-blind, Randomized, Controlled, Factorial 2x2 Trial ("OMEGA3" Study)
Brief Title: Effects of n3 LC PUFAs on Inflammatory, Immune and Senescence Features in Polyvascular Older Subjects (OMSAGE)
Acronym: OMSAGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Collaborators: University of Mons (Other); Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Korpak Kéziah, Korpak Kéziah, medical doctor, Université Libre de Bruxelles
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: B4062021000187
Record Dates: First submitted 2024-10-24; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Polyvascular Disease
Keywords: fatty acid, omega 3; immune response; inflammatory mediators; macrophage polarisation

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, double-blind, 2x2 factorial study among polyvascular subjects over 75 years of age (presence of two or more clinical locations of atherosclerosis) Patients were defined as having polyvascular disease in cases of vascular lesions in ≥2 disease territories or any combination of coronary, peripheral, or carotid artery disease according to the ROCKET AF trial. Coronary artery disease was defined as a history of percutaneous coronary intervention, myocardial infarction, or coronary artery bypass graft surgery. Peripheral artery disease was defined as intermittent amputation for arterial insufficiency, claudication, or a history of vascular reconstruction or bypass surgery. The presence of carotid stenosis was defined as a history of ≥50% stenosis in at least one carotid artery as defined on any imaging modality.
  A total of 80 participants will be studied (20 participants in each arm)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Olive oil
  Interventions: Dietary Supplement: Placebo
- Predominant EPA (Active Comparator): 4 capsules MorEPA plus (Minami Neslé) daily; 590 mg EPA (20:5 n-3) and 130 mg DHA (22:6 n-3)/gels Total: 2360 mg EPA + 520 mg DHA daily; Total in n-3: 2880 mg daily
  Interventions: Dietary Supplement: Long chain polyunsaturated Omega-3
- Predominant DHA (Active Comparator): 4 capsules MorDHA (Minami Neslé) daily; 480 mg DHA (22:6 n-3) and 104 mg EPA (20:5 n-3)/gels Total: 1920 mg DHA + 416 mg EPA daily; Total in n-3: 2336 mg daily
  Interventions: Dietary Supplement: Long chain polyunsaturated Omega-3
- EPA and DHA combined (Active Comparator): 2 capsules Mor DHA (total 1220 mg DHA) + 2 soft gels Mor EPA (total 1388 mg EPA): 2608 mg daily
  Interventions: Dietary Supplement: Long chain polyunsaturated Omega-3

INTERVENTIONS:
Dietary Supplement: Long chain polyunsaturated Omega-3 — 2 capsules of fatty acids in the morning and 2 capsules in the evening except the first day, 4 soft gels in a single administration in the morning, ± 2,6 g/d
  Arms: EPA and DHA combined; Predominant DHA; Predominant EPA
Dietary Supplement: Placebo — Olive oil
  Arms: Placebo

SUMMARY:
The objectives is to evaluate the effect of omega-3 fatty acids in old participants with polyvascular disease on immune parameters and inflammatory mediators at different times. Three modalities of administration of omega-3 will be compared with a placebo (olive oil): predominant EPA (Eicosapentaenoic acid), predominant DHA (doxosahexaenoic acid), and combinaison of both. This study will measure the level of omega3 fatty acids in this population 4 hours after taking, on the 7th day, on the 21th day of administration and 1 month after administration.

DETAILED DESCRIPTION:
Medical Background

Declines in immune function with age and an imbalance between pro- and anti-inflammatory mechanisms lead to a high incidence of infectious and cardiovascular disease among older individuals. ω-3 polyunsaturated fatty acids (EPA and DHA) are anti-inflammatory and represent a substrate of potent mediators, termed specialized proresolving mediators (SPMs). Specialized proresolving mediators (SPMs) are known to limit excessive neutrophil and monocyte migration and stimulate the uptake of apoptotic neutrophils and microbes, thus promoting the resolution of inflammation. Increases in SPM concentrations are linked with decreased uptake of oxidized low-density lipoproteins . Phagocyte functional decline with senescence has been well established. Aged macrophages exhibit functional changes such as compromised chemotaxis, impaired ability to phagocytose pathogenic bacteria, reduced expression of MHC class II molecules and decreased capacity for antigen presentation. However, how phagocyte dysfunction changes with the acquisition of a senescence phenotype is currently unknown.

Some components, such as polyunsaturated fatty acids (n-3 PUFAs), also prevent the induction of senescence and atherosclerosis but also have extensive immunomodulatory effects. The supplementation of fish oil (4 g n-3 PUFA/d) for 3 weeks in healthy older subjects induced dynamic reshaping of human CD4+ T cells and plasma membrane organization. Additionally, 5 days of n-3 PUFA supplementation was associated with an increase in the phagocytic activity of peripheral blood monocytes and neutrophils. The utility of n-3 PUFA-enriched supplements in the prevention of cardiovascular disease has been highlighted. Recently, the EVAPORATE study revealed that the combination of icosapentethyl, a highly purified form of eicopentaenoic acid ethyl ester, and statins might increase the regression of low-attenuation plaque volume on multidetector computed tomography compared with a placebo over 18 months. Specialized proresolving mediators (SPMs), bioactive lipids derived from n-3 PUFAs and leading to the resolution of inflammation, seem to be potential biomarkers for determining the immune regulatory potential of n-3 PUFAs. While native and mox LDL induce the release of inflammatory cytokines and mediators derived from docosahexaenoic acid (DHA) resolvin D1 from young endothelial cells, the effect of mox-LDL in senescent cells on SPM production is unknown. Eicosapentaenoic acid (EPA) and DHA significantly reduce H2O2-induced senescence-associated β-galactosidase activity in cells (by 31% and 22%, respectively). The consumption of fish oil, the main source of n-3 PUFAs, increases phagocytosis and the population of CD4+ and CD8+ lymphocytes in forty-five older healthy Caucasian women.

Drug profile

The substances evaluated will be polyunsaturated fatty acids such as eicosapentaenoic acid (EPA or C20: 5ω-3) and docosahexaenoic acid (DHA or C22: 6 ω-3).

EPA and DHA are known for their anti-inflammatory effects through the inhibition of NFkB pathway activation, the decrease in lipid raft formation, entry into competition with arachidonic acid and the formation of lower-intensity eicosanoids and leukotrienes. They are also known to generate proresolutive mediators called SPMs, such as resolvins, protectins, and maresins. Although their effects are anti-inflammatory and proresolutive, they do not present immunosuppressive effects. The impact of these molecules on different endpoints and on different populations seems less obvious. People with vascular disease may be more sensitive to the effects of these molecules.

Rationale

Study population - dose-duration-administration schedule and hypothesis

Omega-3 fatty acids are important structural components of cell membranes and contribute to various membrane functions, such as fluidity, permeability, the activity of membrane-bound enzymes and receptors, and signal transduction. In 2006, Rees et al reported that 60-year-old subjects were more sensitive to the immunologic effects of EPA and that the neutrophil respiratory burst was lower in those with EPA intake greater than 2,7 g/day. Additionally, the most notable cellular and biochemical changes reported in a study conducted by Schaller et al. occurred in 70-year-old patients with peripheral artery disease. Supplementation for 5 days led to an increase in the phagocytic activity of peripheral blood monocytes and neutrophils. Immunonutrition containing more than 2 g/day of omega-3 has shown encouraging preventive effects against infectious postoperative complications among 65-year-old subjects. The duration of drug administration was only 5 consecutive days. The investiguators hypothesize that a dose of ± 2 g per day for 7 days among older subjects with vascular disease will be sufficient to affect monocyte function (macrophage polarisation) and lymphocyte function after 21 days. The investiguators also propose that a combination of DHA at a lower dose combined with EPA will have the same or a better effect on immune parameters than EPA or DHA alone. A eventual"residual effect" observed 30 days after the last administration will be measured.

The investiguators suggest that of atherosclerotic lesions in older individuals induce high-level secretory components, known as the senescence-associated secretory phenotype (SASP), and induce insufficient proresolutive responses in peripheral blood mononuclear cells, which can be reversed by EPA and DHA in different ways. The investiguators aimed to observe the effects of LC n-3 PUFAs on immune cells through improvements in inflammatory and senescence markers.

Design

This monocentric study is an interventional experimental plan to understand physiopathological processes in older subjects. This randomized, controlled, double-blind, 2x2 factorial trial will be performed in polyvascular subjects over 75 years of age, without direct individual benefit.

A total of 80 participants (20 participants in each arm) were divided into 4 groups. One group will receive ± 2,4 g/day of DHA, a second will receive ± 2,4 g/d of EPA, and a third group will receive a combination of DHA and EPA. The control group will receive a placebo.

To respect the blindness procedure (double-blind), the total number of capsules to be taken by the patient per day will be 2 capsules in the morning and 2 capsules in the evening for 21 days. On the first day and in the morning, the subject took all 4 capsules at one time.

Biological parameters will be measured prospectively from blood samples taken at different times. Each subject will end his participation on the 51st day, the day of the last visit, with a blood test.

Block randomization will be performed and stratified by sex.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 75 years old
* Patients with polyvascular disease in cases of vascular lesions in ≥2 disease territories or any combination of coronary, peripheral, or carotid artery disease.
* Able to comply with the requirements of the study protocol
* Signed informed consent form approved by the ethical committee
* No illness or event within 2 months prior to inclusion (hospitalization, trauma, active cancer, infection, acute failure of chronic disease, surgical intervention)
* No history of multiple and/or severe allergies to drugs or foods
* No consumption of fish oil or omega-3 fatty acid supplements within 2 months prior to inclusion
* No consumption of more than 500 mg/day of dietary omega-3 fatty acids (questionnaire)
* No intake of anti-inflammatory or corticosteroid medication within 2 weeks prior to inclusion
* Able and authorized to take a pill
* No intervention planned in the months following the start of the study

Exclusion Criteria:

* Inflammatory syndrome (CRP >10 mg/l) on day 0 and day 7
* Acute illness or event during the time of intervention

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-11-04 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Attenuation of production of inflammatory mediators | Day 0, Day 21
  lowering plasma IL8 in pg/ml

SECONDARY OUTCOMES:
Enhanced production of proresolving mediators | Day 0, Day 21
  Production of plasma proresolving mediators (plasma RvD1, RvE1, 17-HDHA, 18-HEPE LTB4 level in pg/ml plasma)
Increased level of EPA and DHA | Day 0, 4 hours post dose , Day 7, Day 21, Day 56
  To measure the level of omega-3 in this population 4 hours after consumption (kinetics), on the 7th day of administration, on the 21st day and 1 month after administration (plasma EPA, DHA and AA level in pg/ml) and improved Omega6/3 ratio
Attenuation of production of senescence-associated secretory phenotype | Day 0, Day 21
  lowering level of supernatant IL8 in pg/mL after incubation of serum with endothelial cells
Attenuation of production of inflammatory mediators from immune cells | Day 0, Day 21
  Lowering level of supernatant IL8 in pg/mL after stimulation of macrophage by calcium ionophore
Improving immune parameters | Day 0, Day 7, Day 21, Day 51
  Lowering intermediate and non-classical M2 monocytes subsets in percent

OTHER OUTCOMES:
Lowering features of senescence | Day 0, Day 21
  Lowering marker senescence associated-β-galactosidase (SAβgal) mesured in % of activity on endothelial cells after incubation of serum

CONTACTS AND LOCATIONS:
Overall Officials: Karim Zouaoui Boudjeltia, PhD, Study Director — Laboratory of Experimental Medicine

IPD SHARING:
Plan to Share IPD: No
This access was not discussed with the ethics committees for approval